CLINICAL TRIAL: NCT02072915
Title: Randomized Single Blind Controlled Trial of EUS-FNA With and Without Suction for Adequate Cellblock Sample Procurement of Solid Pancreatic Mass Lesions Using 25G Needle
Brief Title: EUS-FNA With and Without Suction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: F131108005
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Solid Pancreatic Mass Lesions
MeSH Terms: interventions — Suction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suction (Experimental): Suction will be applied to patients undergoing EUS-FNA
  Interventions: Procedure: Suction
- Without suction (No Intervention): No suction will be applied to patients undergoing EUS-FNA

INTERVENTIONS:
Procedure: Suction
  Arms: Suction

SUMMARY:
To compare the number of passes required for cellblock acquisition with and without suction using the 25g needle.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to UAB Endoscopy Unit for assessment of pancreatic mass lesions that requires FNA.

Exclusion Criteria:

* Age < 19 years

  * Unable to safely undergo EUS for any reason
  * Coagulopathy (INR>1.6, Prothrombin Time>18 secs, Thrombocytopenia < 80,000 cells/ml)
  * Unable to consent
  * Non-English speaking patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of passes | once at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jayapal Ramesh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States